CLINICAL TRIAL: NCT03227237
Title: Assess the Impact of Strained Interpersonal Relationship (IPR) With Parents on Juvenile Delinquency Among Children Residing in Selected Delinquent Home Ambala, Haryana"
Brief Title: Impact of Strained Interpersonal Relationship (IPR) With Parents on Juvenile Delinquency Among Children
Status: Completed | Type: Observational
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Talwinder Kaur, M.Sc Nursing, Maharishi Markendeswar University (Deemed to be University)
Other Study IDs: 788
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Interpersonal Relations
Keywords: Impact, Interpersonal Relationship, Juvenile delinquency
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Introduction was given about research and researcher to participants. Got the assent from participants, consent from parents and collected baseline data (demographic variable, specific IPR variable) from the participants. Collected data about IPR on the basis of Modified Washington State Juvenile Court Assessment Scale from the participants.Participants were asked to fill out IPR related information of pre delinquent period with paper & pencil mode of technique. It took for each group of participants about 40 minutes. Collected data regarding conduct variables from parents with interview technique. On each day 8-16 participants were covered.
- Control group: Introduction was given about research and researcher to participants. Confirmed telephonic consent from Parents.Collected baseline data (demographic variable, specific IPR variable) from the participants.Collected data about IPR on the basis of Modified Washington State Juvenile Court Assessment Scale from the participants. Participants were asked to fill out IPR related information of their past life from before 2 years with paper & pencil mode of technique. It took for each group of participants about 40 minutes. On each day 8-20 participants were covered Got the written consent form parents and collected data regarding conduct variables from parents with interview technique.

SUMMARY:
"Assess the impact of Strained Interpersonal Relationship (IPR) with parents on Juvenile Delinquency among Children residing in Selected Delinquent Home Ambala, Haryana"

DETAILED DESCRIPTION:
The objectives of this study are:- To assess and compare IPR score with parents among case (delinquent children) and control (non delinquent children) group.

To determine the association of IPR score with selected variables among case (delinquent children) and control (non delinquent children) group.

ELIGIBILITY:
Inclusion Criteria:

children who were aged 13-18 years and residing in selected delinquent home, ambala (for case).

aged 13- 18 years, fulfils matching (age) and homogenity(gender) with case and studing in selected school, Barara (for control).

alert, oriented and able to read, comprehend and speak English/ hindi.

Exclusion Criteria:

children who were non-literate (for case) not willing to participate in study. not having both biological parents.

Ages: 13 Years to 18 Years | Sex: Male
Age Groups: Child, Adult
Gender Based: Yes — Male with age of 13-18 years
Study Population: The sample in the present study is Delinquent Children(case) in Govt. Delinquent Home, Ambala and Non Delinquent children (control) in Govt. Senior Secondary school of Barara, Haryana. sampling technique used was Total enumerative sampling for case group and convenience sampling based on matching (age) and homogenity (gender) for control group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Interpersonal Relation | 40 minutes per group
  The IPR score was categorized into three categories, Very poor IPR (26-51), Poor IPR (52-64), and Good IPR with parents (65-78)

CONTACTS AND LOCATIONS:
Overall Officials: Talwinder Kaur, Master, Principal Investigator — Maharishi Markandeshwar University
Locations (1):
- Talwinder kaur, Yamuna Nagar, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrenkohl TI, Maguin E, Hill KG, Hawkins JD, Abbott RD, Catalano RF. Developmental risk factors for youth violence. J Adolesc Health. 2000 Mar;26(3):176-86. doi: 10.1016/s1054-139x(99)00065-8. PMID 10706165
- [Background] Mednick BR, Baker RL, Carothers LE. Patterns of family instability and crime: The association of timing of the family's disruption with subsequent adolescent and young adult criminality. J Youth Adolesc. 1990 Jun;19(3):201-20. doi: 10.1007/BF01537887. PMID 24272449
- [Background] Hoeve M, Stams GJ, van der Put CE, Dubas JS, van der Laan PH, Gerris JR. A meta-analysis of attachment to parents and delinquency. J Abnorm Child Psychol. 2012 Jul;40(5):771-85. doi: 10.1007/s10802-011-9608-1. PMID 22278802